CLINICAL TRIAL: NCT00750464
Title: Collection of Raw Data of Thermal Imaging for the Purpose of Developing a Device for Early Detection of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Real Imaging Ltd. (Industry)
Responsible Party: Mr. Boaz Arnon, CEO, Real Imaging Ltd.
Other Study IDs: Pr-118-8061 ver. 001
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Collection of thermal "images" of women with breast tumors in varying degrees of severity in order to evaluate and improve Real Imaging's device ("RI3.0") capabilities , which will assist in early detection of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a breast abnormality (identified by mammography, ultrasound, MRI and/or a clinical examination) requiring a biopsy.

Exclusion Criteria:

* Subjects who have had a mammography, ultrasound, and/or MRI examination performed on the day of the study, prior to being "imaged" by RI3.0.
* Subjects who have undergone any type of breast surgery throughout the 6 weeks preceding the study.
* Subjects who have had a breast biopsy performed throughout the 6 weeks preceding the study.
* Subjects who have undergone a mastectomy.
* Subjects who have a large scar (causing breast deformation) following breast lumpectomy and/or any other cause (e.g. accident).
* Subjects with prior breast reduction surgery or breast augmentation surgery.
* Subjects who have a fever on the day of their biopsy.
* Subjects who are pregnant.
* Subjects who are breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a breast abnormality (identified by mammography, ultrasound, MRI and/or a clinical examination) requiring a biopsy
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2008-11; Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miri Sklair-Levy, MD, Principal Investigator — Hadassah Medical Organization, Jerusalem
Locations (4):
- Israel (4):
  - Carmel Medical Center - Lin, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva